CLINICAL TRIAL: NCT03483584
Title: A Prospective Longitudinal Cohort Study to Determine the Incidence of HIV-associated Non-AIDS Conditions in Newly Diagnosed HIV-infected Individuals Initiating Integrase Inhibitor-based and Other Anti-retroviral Regimens
Brief Title: Incidence of HANA Conditions in HIV-infected Individuals
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Grace Lui, Clinical Assistant Professor, Chinese University of Hong Kong
Other Study IDs: HANA protocol v.1 10Oct2017
Record Dates: First submitted 2018-03-25; First posted 2018-03-30 (Actual); Results first posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: HIV; Metabolic Syndrome; Osteopenia; Osteoporosis; Vitamin D Deficiency; Renal Impairment; Liver Fibroses
MeSH Terms: conditions — Metabolic Syndrome; Bone Diseases, Metabolic; Osteoporosis; Vitamin D Deficiency; Renal Insufficiency; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- INSTI: INSTI-containing ART regimens
- non-INSTI: non-INSTI-containing ART regimens

SUMMARY:
With the availability of effective anti-retroviral therapy, HIV-infected individuals are expected not to die of AIDS and have longer life expectancy. But at the same time, HIV-associated non-AIDS (HANA) conditions are becoming more important in their clinical management. It is currently uncertain whether patients started on different anti-retroviral regimens will have different incidence of HANA conditions.

This study aims to evaluate the incidence of various HANA conditions in a cohort of newly diagnosed HIV-infected individuals in Hong Kong initiating anti-retroviral treatment. The incidence of various HANA conditions will be evaluated for those receiving INSTI versus other non-INSTI-based regimens.

The HANA conditions evaluated will include 1. Hypertension 2. Diabetes and insulin resistance 3. Dyslipidemia 4. Lipodystrophy 5. Metabolic syndrome 6. Osteopenia and osteoporosis 7. Vitamin D deficiency 8. Renal impairment and kidney tubular dysfunction and 9. Liver fibrosis. Patients will be assessed prior to initiation of anti-retroviral therapy, and 48 weeks and 96 weeks after initiation of treatment. The incidence of development of each HANA condition will be determined and compared between those initiated different anti-retroviral regimens.

DETAILED DESCRIPTION:
This is a prospective, longitudinal, cohort study. 150 newly diagnosed HIV-infected individuals attending HIV clinics in Hong Kong will be recruited. Clinical assessment, and laboratory and imaging studies will be performed at baseline prior to initiation of anti-retroviral regimen, then annually thereafter for 5 years. Choice of anti-retroviral regimen will be decided by the in-charge HIV physician. Incidence of development of various HANA will be determined in those initiated INSTI-based regimens and other anti-retroviral regimens. An electronic platform will be used to formulate risk prediction for various clinical outcomes, and serve as a clinical decision support tool.

Statistical analysis;

1. The incidence rate of each HANA defined as above will be calculated as:
2. The incidence rate of each HANA will be determined for subjects started INSTI-based regimens and other non-INSTI-anti-retroviral regimens.
3. Variables, including demographic, clinical, treatment-related, and laboratory parameters, will be evaluated for association with development of various HANA, in univariate and multivariate analyses. Analyses will be performed for the whole cohort, and subgroup analyses will be performed in those initiated INSTI-based regimens and other non-INSTI-based regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed HIV infection by HIV antibody or RNA test
2. Age ≥18 years old
3. Anti-retroviral treatment naïve
4. Agree to initiate anti-retroviral therapy (ART) as determined by in-charge HIV physician

Exclusion Criteria:

1. Pregnancy
2. Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All newly diagnosed HIV-infected patients meeting inclusion criteria, who attend the government HIV clinic, which is the largest HIV clinic in Hong Kong, over a 12-month period, will be invited to participate in this study. Subjects will also be referred by non-governmental organizations providing support to HIV-infected individuals at the time of diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace Lui, Principal Investigator — CUHK
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During the study period, a prospective and longitudinal cohort study involving People living with HIV (PLWH) recruited from the Infectious Diseases Clinic of the Prince of Wales Hospital, Hong Kong SAR, from April 2018 to May 2022. PLWH initiating or switching to a new ART regimen within 6 months were enrolled. Participants were assessed at baseline and followed up annually for 2 years to assess for the presence of various HANA conditions.
Groups:
- INSTI: Participants on INSTI-based antiretroviral therapy at baseline
- non-INSTI: Participants on non-INSTI-based antiretroviral therapy at baseline
Period: Overall Study
Arm/Group | INSTI | non-INSTI
Started (Participants eligible to the study were enrolled to the study.) | 183 | 32
At year 1 (Participants had follow-up study visits at year 1) | 131 | 22
At year 2 (Participants had follow-up study visits at year 2) | 110 | 21
Completed (Only participants who had baseline and at least one follow-up visits during the two-year follow-up period were included in the data analysis.) | 139 | 24
Not Completed | 44 | 8
Not completed — Lost to Follow-up | 40 | 7
Not completed — Withdrawal by Subject | 4 | 1

BASELINE CHARACTERISTICS:
Population: 215 participants were recruited into the study. Those participants who had baseline and at least one follow-up visit during the two-year follow-up period were included in the data analyses. Those who had only one study visits were excluded from final analyses.
Groups:
- INSTI: INSTI-based antiretroviral therapy
- Non-INSTI: non-INSTI-based antiretroviral therapy
- Total: Total of all reporting groups
Arm/Group | INSTI | Non-INSTI | Total
Number analyzed (Participants) | 183 | 32 | 215
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (14.5) | 48.8 (12.7) | 46.7 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 4 | 27
  Male | 160 | 28 | 188
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 174 | 30 | 204
  Non-Chinese | 9 | 2 | 11
Duration of HIV diagnosis [Median (Inter-Quartile Range); unit: years] | 0.8 [0.2 to 8.4] | 7.7 [0.5 to 14.0] | 1.0 [0.2 to 9.6]

OUTCOME MEASURES:

1. Primary Outcome: Prevalences of HIV-associated Non-AIDS Conditions (HANA)
Description: Participants who were assessed at baseline and at least one of follow-up visits were included in the data analysis for prevalence of HIV-associated non-AIDS conditions (HANA)
  Prevalences of the following HIV-associated non-AIDS conditions (HANA) were assessed at baseline.
  * hypertension
  * diabetes mellitus
  * insulin resistance
  * dyslipidemia
  * metabolic syndrome
  * osteoporosis
  * osteopenia
  * vitamin D deficiency
  * renal disease
  * kidney tubular dysfunction
  * intermediate or advanced fibrosis (FIB-4 >1.3)
  * advanced fibrosis (FIB-4 >2.67)
Time Frame: Baseline
Population: Participants who had baseline and at least one follow-up study visits were included in the analyses.
Measure: Count of Participants; unit: Participants
Groups:
- non-INSTI: non-INSTI based antiretroviral therapy
Arm/Group | INSTI | non-INSTI
Number analyzed (Participants) | 139 | 24
Participants
  Prevalence of hypertension | 69 | 15
  Prevalence of diabetes mellitus | 30 | 4
  Prevalence of insulin resistance | 79 | 9
  Prevalence of dyslipidemia | 85 | 17
  Prevalence of metabolic syndrome | 60 | 16
  Prevalence of osteopenia | 72 | 9
  Prevalence of osteoporosis | 6 | 1
  Prevalence of vitamin D deficiency | 27 | 3
  Prevalence of renal diseases | 58 | 9
  Prevalence of kidney tubular dysfunction | 55 | 9
  Prevalence of intermediate or advanced fibrosis (FIB-4 >1.3) | 42 | 10
  Prevalence of advanced fibrosis (FIB-4 >2.67) | 5 | 1
Statistical Analysis 1: Comparison: INSTI vs non-INSTI; Test type: Other — Chi-square test is to detect the difference in the prevalence of hypertension between INSTI and non-INSTI groups; p = 0.244, Chi-squared — The threshold for significance was set at p < 0.05
Statistical Analysis 2: Comparison: INSTI vs non-INSTI; Test type: Other — Chi square test is to detect the difference in prevalence of diabetes mellitus between INSTI and non-INSTI groups; p = 0.584, Chi-squared — The threshold for significance was set at p < 0.05
Statistical Analysis 3: Comparison: INSTI vs non-INSTI; Test type: Other — Chi square test is used to detect the difference in prevalence of insulin resistance between INSTI and non-INSTI groups; p = 0.067, Chi-squared — The threshold for significance was set at p < 0.05
Statistical Analysis 4: Comparison: INSTI vs non-INSTI; Test type: Other — Chi square test is used to detect the difference in prevalence of dyslipidemia between INSTI and non-INSTI groups; p = 0.365, Chi-squared — The threshold for significance was set at p < 0.05
Statistical Analysis 5: Comparison: INSTI vs non-INSTI; Test type: Other — Chi square test is used to detect the difference in prevalence of metabolic syndrome between INSTI and non-INSTI groups; p = 0.033, Chi-squared — The threshold for significance was set at p < 0.05
Statistical Analysis 6: Comparison: INSTI vs non-INSTI; Test type: Other — Chi square is used to detect the difference in prevalence of osteopenia between INSTI and non-INSTI groups; p = 0.196, Chi-squared — The threshold for significance was set at p < 0.05
Statistical Analysis 7: Comparison: INSTI vs non-INSTI; Chi square test is used to detect the difference in prevalence of osteoporosis between INSTI and non-INSTI groups; Test type: Other; p = 1.000, Fisher Exact — The threshold for significance was set at p < 0.05; Fisher exact test is used when any cells have expected count less than 5
Statistical Analysis 8: Comparison: INSTI vs non-INSTI; Chi square test is used to detect the difference in prevalence of vitamin D deficiency between INSTI and non-INSTI groups; Test type: Other; p = 0.572, Fisher Exact — The threshold for significance was set at p < 0.05; Fisher exact test is used when any cells have expected less than 5
Statistical Analysis 9: Comparison: INSTI vs non-INSTI; Chi square test is used to detect the difference in prevalence in renal disease between INSTI and non-INSTI groups; Test type: Other; p = 0.698, Chi-squared — The threshold for significance was set at p < 0.05
Statistical Analysis 10: Comparison: INSTI vs non-INSTI; Test type: Other — Chi square test is used to detect the difference in prevalence of kidney tubular dysfunction between INSTI and non-INSTI groups; p = 0.848, Chi-squared — The threshold for significance was set at p < 0.05
Statistical Analysis 11: Comparison: INSTI vs non-INSTI; Test type: Other — Chi square test is used to detect the difference in prevalence of intermediate or advanced fibrosis (FIB-4 >1.3) between INSTI and non-INSTI groups; p = 0.274, Chi-squared — The threshold for significance was set at p < 0.05
Statistical Analysis 12: Comparison: INSTI vs non-INSTI; Test type: Other — Chi square test is used to detect the difference in prevalence of advanced fibrosis (FIB-4 >2.67) between INSTI and non-INSTI groups; p = 1.000, Fisher Exact — The threshold for significance was set at p < 0.05; Fisher exact test is used when any cells have expected count less than 5

2. Primary Outcome: Incidence Rates of HANA Conditions for At-risk Groups
Description: Participants who were assessed at baseline and at least one of follow-up visits were included in the data analysis for incidence rates of HANA
  Incidence rates of following HANA conditions were reported among at-risk INSTI and non-INSTI-based antiretroviral therapy at 2 years.
  * hypertension
  * diabetes mellitus
  * insulin resistance
  * dyslipidemia
  * metabolic syndrome
  * osteopenia
  * osteoporosis
  * vitamin D deficiency
  * renal disease
  * kidney tubular dysfunction
  * intermediate or advanced fibrosis (FIB-4 > 1.3)
  * advanced fibrosis (FIB-4 >2.67)
Time Frame: Enrollment to 2 years
Population: At risk participants who had baseline and at least one follow-up study visits during the two-year period were included in the analysis. Incidence rates of HANA-conditions were reported in INSTI and non-INSTI groups. A person-year is a unit expressing the cumulative observation time during which the population is at risk for HANA conditions. Incidence rates are expressed as the number of new cases developing HANA conditions per 100 at-risk person-years during the study period.
Measure: Number (95% Confidence Interval); unit: cases per 100-persons years
Arm/Group | INSTI | non-INSTI
Number analyzed (Participants) | 139 | 24
cases per 100-persons years
  Incidence rates of hypertension: number analyzed (Participants) | 70 | 9
  Incidence rates of hypertension | 14.7 [9.5 to 22.8] | 10.5 [2.6 to 42.1]
  Incidence rate of diabetes mellitus: number analyzed (Participants) | 109 | 20
  Incidence rate of diabetes mellitus | 3.3 [1.6 to 6.9] | 9.5 [3.6 to 25.4]
  Incidence rates of insulin resistance: number analyzed (Participants) | 58 | 15
  Incidence rates of insulin resistance | 31.6 [22.9 to 43.6] | 41.9 [24.4 to 72.2]
  Incidence rates of dyslipidemia: number analyzed (Participants) | 54 | 7
  Incidence rates of dyslipidemia | 16.5 [10.3 to 26.6] | 14.3 [3.6 to 57.1]
  Incidence rates of metabolic syndrome: number analyzed (Participants) | 79 | 8
  Incidence rates of metabolic syndrome | 9.9 [5.9 to 16.4] | 11.8 [2.9 to 47.0]
  Incidence rates of osteopenia: number analyzed (Participants) | 67 | 15
  Incidence rates of osteopenia | 5.1 [2.4 to 10.7] | 3.4 [0.5 to 24.5]
  Incidence rates of osteoporosis: number analyzed (Participants) | 133 | 23
  Incidence rates of osteoporosis | 1.1 [0.4 to 3.5] | 0 [0 to 0]
  Incidence rates of vitamin D deficiency: number analyzed (Participants) | 110 | 21
  Incidence rates of vitamin D deficiency | 16.7 [12.1 to 22.9] | 7.1 [2.3 to 22.1]
  Incidence rates of renal diseases: number analyzed (Participants) | 81 | 15
  Incidence rates of renal diseases | 20.1 [14.2 to 28.6] | 17.2 [7.2 to 41.4]
  Incidence rates of kidney tubular dysfunction: number analyzed (Participants) | 84 | 15
  Incidence rates of kidney tubular dysfunction | 16.3 [11.2 to 23.9] | 13.3 [5.0 to 35.3]
  Incidence rates of intermediate or advanced fibrosis (FIB-4 >1.3): number analyzed (Participants) | 90 | 13
  Incidence rates of intermediate or advanced fibrosis (FIB-4 >1.3) | 6.7 [3.8 to 11.8] | 11.5 [3.7 to 35.8]
  Incidence rates of advanced fibrosis (FIB-4 >2.67): number analyzed (Participants) | 127 | 22
  Incidence rates of advanced fibrosis (FIB-4 >2.67) | 1.9 [0.8 to 4.6] | 0 [0 to 0]
Statistical Analysis 1: Comparison: INSTI vs non-INSTI; Crude incidence rate ratio (IRR) was expressed as a ratio of incidence rates of developing hypertension in INSTI group compared with non-INSTI group as reference group at 2 years; Test type: Other — Poisson loglinear; Incidence rate ratio = 1.508, 95% CI 2-sided [0.352 to 6.450] — Wald chi square test is used to investigate whether INSTI group had a higher risk of developing of HANA conditions compared with non-INSTI group, with IRR >1 meaning higher risk of developing new HANA conditions
Statistical Analysis 2: Comparison: INSTI vs non-INSTI; Adjusted Incidence rate ratio (IRR) was expressed as a ratio of incidence rate of developing hypertension in INSTI group compared with non-INSTI group at 2 years after adjusted by age, sex, treatment-naive or experienced, duration of HIV diagnosis, baseline body weight and CD4 count; Test type: Other — Poisson loglinear; Incidence rate ratio = 1.936, 95% CI 2-sided [0.251 to 14.919] — Wald chi square test is used to detect the difference in incidence rates in the INSTI group compared with the non-INSTI group (as reference group) after adjustment of covariates, with IRR >1 meaning higher risk of developing new HANA conditions
Statistical Analysis 3: Comparison: INSTI vs non-INSTI; Crude incidence rate ratio (IRR) was expressed as a ratio of incidence rates of developing diabetes mellitus in INSTI group compared with non-INSTI group as reference group at 2 years; Test type: Other — Poisson loglinear; Incidence rate ratio = 0.388, 95% CI 2-sided [0.099 to 1.155] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: INSTI vs non-INSTI; Adjusted Incidence rate ratio (IRR) was expressed as a ratio of incidence rate of developing diabetes mellitus in INSTI group compared with non-INSTI group at 2 years after adjusted by age, sex, treatment-naive or experienced, duration of HIV diagnosis, baseline body weight and CD4 count; Test type: Other — Poisson loglinear; Incidence rate ratio = 0.507, 95% CI 2-sided [0.132 to 1.948] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 5: Comparison: INSTI vs non-INSTI; Crude incidence rate ratio (IRR) was expressed as a ratio of incidence rates of developing insulin resistance in INSTI group compared with non-INSTI group as reference group at 2 years; Test type: Other — Poisson loglinear; Incidence rate ratio = 0.743, 95% CI 2-sided [0.395 to 1.397] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: INSTI vs non-INSTI; Adjusted Incidence rate ratio (IRR) was expressed as a ratio of incidence rate of developing insulin resistance in INSTI group compared with non-INSTI group at 2 years after adjusted by age, sex, treatment-naive or experienced, duration of HIV diagnosis, baseline body weight and CD4 count; Test type: Other — Poisson loglinear; Incidence rate ratio = 0.883, 95% CI 2-sided [0.444 to 1.759] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 7: Comparison: INSTI vs non-INSTI; Crude incidence rate ratio (IRR) was expressed as a ratio of incidence rates of developing dyslipidemia in INSTI group compared with non-INSTI group as reference group at 2 years; Test type: Other — Poisson loglinear; Incidence rate ratio = 1.187, 95% CI 2-sided [0.274 to 5.139] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: INSTI vs non-INSTI; Adjusted Incidence rate ratio (IRR) was expressed as a ratio of incidence rate of developing dyslipidemia in INSTI group compared with non-INSTI group at 2 years after adjusted by age, sex, treatment-naive or experienced, duration of HIV diagnosis, baseline body weight and CD4 count; Test type: Other — Poisson loglinear; Incidence rate ratio = 1.210, 95% CI 2-sided [0.257 to 5.688] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 9: Comparison: INSTI vs non-INSTI; Crude incidence rate ratio (IRR) was expressed as a ratio of incidence rates of developing metabolic syndrome in INSTI group compared with non-INSTI group as reference group at 2 years; Test type: Other — Poisson loglinear; Incidence rate ratio = 0.855, 95% CI 2-sided [0.196 to 3.739] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: INSTI vs non-INSTI; Adjusted Incidence rate ratio (IRR) was expressed as a ratio of incidence rate of developing metabolic syndrome in INSTI group compared with non-INSTI group at 2 years after adjusted by age, sex, treatment-naive or experienced, duration of HIV diagnosis, baseline body weight and CD4 count; Test type: Other — Poisson loglinear; Incidence rate ratio = 0.534, 95% CI 2-sided [0.108 to 2.631] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 11: Comparison: INSTI vs non-INSTI; Crude incidence rate ratio (IRR) was expressed as a ratio of incidence rates of developing osteopenia in INSTI group compared with non-INSTI group as reference group at 2 years; Test type: Other — Poisson loglinear; Incidence rate ratio = 1.396, 95% CI 2-sided [0.172 to 11.350] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 12: Comparison: INSTI vs non-INSTI; Adjusted Incidence rate ratio (IRR) was expressed as a ratio of incidence rate of developing osteopenia in INSTI group compared with non-INSTI group at 2 years after adjusted by age, sex, treatment-naive or experienced, duration of HIV diagnosis, baseline body weight and CD4 count; Test type: Other — Poisson loglinear; Incidence rate ratio = 1.053, 95% CI 2-sided [0.119 to 9.317] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 13: Comparison: INSTI vs non-INSTI; Crude incidence rate ratio (IRR) was expressed as a ratio of incidence rates of developing osteoporosis in INSTI group compared with non-INSTI group as reference group at 2 years; Test type: Other — Poisson loglinear; Incidence rate ratio = 0, 95% CI 2-sided [0 to 0] — No incidence of osteoporosis was reported in non-INSTI group at 2 years
Statistical Analysis 14: Comparison: INSTI vs non-INSTI; Adjusted Incidence rate ratio (IRR) was expressed as a ratio of incidence rate of developing osteoporosis in INSTI group compared with non-INSTI group at 2 years after adjusted by age, sex, treatment-naive or experienced, duration of HIV diagnosis, baseline body weight and CD4 count; Test type: Other — Poisson loglinear; Incidence rate ratio = 0, 95% CI 2-sided [0 to 0] — No incidence of osteoporosis was reported in non-INSTI group at 2 years
Statistical Analysis 15: Comparison: INSTI vs non-INSTI; Crude incidence rate ratio (IRR) was expressed as a ratio of incidence rates of developing vitamin D deficiency in INSTI group compared with non-INSTI group as reference group at 2 years; Test type: Other — Poisson loglinear; Incidence rate ratio = 2.198, 95% CI 2-sided [0.679 to 7.122] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 16: Comparison: INSTI vs non-INSTI; Adjusted Incidence rate ratio (IRR) was expressed as a ratio of incidence rate of developing vitamin D deficiency in INSTI group compared with non-INSTI group at 2 years after adjusted by age, sex, treatment-naive or experienced, duration of HIV diagnosis, baseline body weight and CD4 count; Test type: Other — Poisson loglinear; Incidence rate ratio = 3.551, 95% CI 2-sided [0.850 to 14.833] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 17: Comparison: INSTI vs non-INSTI; Crude incidence rate ratio (IRR) was expressed as a ratio of incidence rates of developing renal diseases in INSTI group compared with non-INSTI group as reference group at 2 years; Test type: Other — Poisson loglinear; Incidence rate ratio = 1.197, 95% CI 2-sided [0.465 to 3.077] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 18: Comparison: INSTI vs non-INSTI; Adjusted Incidence rate ratio (IRR) was expressed as a ratio of incidence rate of developing renal diseases in INSTI group compared with non-INSTI group at 2 years after adjusted by age, sex, treatment-naive or experienced, duration of HIV diagnosis, baseline body weight and CD4 count; Test type: Other — Poisson loglinear; Incidence rate ratio = 1.538, 95% CI 2-sided [0.510 to 4.638] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 19: Comparison: INSTI vs non-INSTI; Crude incidence rate ratio (IRR) was expressed as a ratio of incidence rates of developing kidney tubular dysfunction in INSTI group compared with non-INSTI group as reference group at 2 years; Test type: Other — Poisson loglinear; Incidence rate ratio = 1.166, 95% CI 2-sided [0.408 to 3.331] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 20: Comparison: INSTI vs non-INSTI; Adjusted Incidence rate ratio (IRR) was expressed as a ratio of incidence rate of developing kidney tubular dysfunction in INSTI group compared with non-INSTI group at 2 years after adjusted by age, sex, treatment-naive or experienced, duration of HIV diagnosis, baseline body weight and CD4 count; Test type: Other — Poisson loglinear; Incidence rate ratio = 2.101, 95% CI 2-sided [0.615 to 7.180] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 21: Comparison: INSTI vs non-INSTI; Crude incidence rate ratio (IRR) was expressed as a ratio of incidence rates of developing intermediate or advanced fibrosis (FIB-4 > 1.3) in INSTI group compared with non-INSTI group as reference group at 2 years; Test type: Other — Poisson loglinear; Incidence rate ratio = 0.563, 95% CI 2-sided [0.159 to 1.995] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 22: Comparison: INSTI vs non-INSTI; Adjusted Incidence rate ratio (IRR) was expressed as a ratio of incidence rate of developing intermediate or advanced fibrosis (FIB-4 > 1.3) in INSTI group compared with non-INSTI group at 2 years after adjusted by age, sex, treatment-naive or experienced, duration of HIV diagnosis, baseline body weight and CD4 count; Test type: Other — Poisson loglinear; Incidence rate ratio = 0.922, 95% CI 2-sided [0.244 to 3.493] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 23: Comparison: INSTI vs non-INSTI; Crude incidence rate ratio (IRR) was expressed as a ratio of incidence rates of developing advanced fibrosis (FIB-4 >2.67) in INSTI group compared with non-INSTI group as reference group at 2 years; Test type: Other — Poisson loglinear; Incidence rate ratio = 0, 95% CI 2-sided [0 to 0] — No incidence in advanced fibrosis (FIB-4 >2.67) was reported in non-INSTI group at 2 years
Statistical Analysis 24: Comparison: INSTI vs non-INSTI; Adjusted Incidence rate ratio (IRR) was expressed as a ratio of incidence rate of developing advanced fibrosis (FIB-4 > 2.67) in INSTI group compared with non-INSTI group at 2 years after adjusted by age, sex, treatment-naive or experienced, duration of HIV diagnosis, baseline body weight and CD4 count; Test type: Other — Poisson loglinear; Incidence rate ratio = 0, 95% CI 2-sided [0 to 0] — No incidence in advanced fibrosis (FIB-4 >2.67) was reported in non-INSTI group at 2 years

ADVERSE EVENTS:
Time Frame: At 96 weeks
Arm/Group | INSTI | non-INSTI
All-Cause Mortality (participants affected / at risk) | 0/139 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/139 | 0/24
Other Adverse Events (participants affected / at risk) | 0/139 | 0/24

LIMITATIONS AND CAVEATS:
Our study was limited by a small sample size, limiting power to compare outcomes between antiretroviral regimens. The study was started before Coronavirus disease 2019 (COVID-19) pandemic, and there were some lost to follow up after baseline visit due to pandemic social measures. The predominance of Asian male participants in this cohort may limit generalizability of the results to other ethnicity and women with HIV.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-05): https://cdn.clinicaltrials.gov/large-docs/84/NCT03483584/Prot_SAP_000.pdf